CLINICAL TRIAL: NCT06799182
Title: The Influence of Periodontal Disease and Periodontal Treatment on Colorectal Cancer
Brief Title: Periodontal Disease and Colorectal Cancer
Acronym: PD and CRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Institute of Oncology Ljubljana (Other); Institute of microbiology and immunology, Slovenia (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120-486/2021/6 PB in KRK
Record Dates: First submitted 2025-01-15; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-11

CONDITIONS: Periodontal Diseases; Colorectal Carcinoma
MeSH Terms: conditions — Periodontal Diseases; Colorectal Neoplasms | interventions — Periodontal Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with colorectal cancer who recived periodontal treatment (Experimental): Patients with colorectal cancer were treated for periodontal disease based on the condition of their periodontal tissues.
  Interventions: Procedure: periodontal treatment
- Patients with colorectal cancer who did not recived periodontal treatment (No Intervention): Due to ethical concerns, we selected patients who had completed cancer therapy before the start of our study for the control group, and who met the inclusion criteria based on the completed questionnaires.

INTERVENTIONS:
Procedure: periodontal treatment — Based on the results of the dental examination and the diagnosis of the periodontal tissue condition according to the new classification of periodontal disease, we performed appropriate non-surgical treatment of periodontal disease, provided oral hygiene instruction, and took a biofilm sample from the deep periodontal pocket. We then collected a sample of the altered mucosa during bowel surgery for colorectal cancer and conducted a microbiological investigation using quantitative culture to compare the presence of Fusobacterium nucleatum and Porphyromonas gingivalis in the pariodontal pocket and altered intestinal mucosa.
  Other Names: Biopsy of the intestinal mucosa for quantitative culture; samples of periodontal biofilm for quantitative culture
  Arms: Patients with colorectal cancer who recived periodontal treatment

SUMMARY:
The aim of this interventional study is to determine the impact of periodontal disease and periodontal treatment on patients with colorectal cancer.

The main questions were:

1. Does periodontal treatment affect the levels of C-reactive protein in the blood of patients undergoing cancer treatment?
2. Can the investigators isolate periodontal pathogenic bacteria Fusobacterium nucleatum and Porphyromonas gingivalis from the mucosa of cancerous colon tissue using the method of quantitative culture?

The investigators will compare the levels of C-reactive protein in the blood of patients undergoing treatment for colorectal cancer who have received periodontal treatment with patients who have not received periodontal treatment. CRP levels will be measured during the first examination with the oncological surgeon, on the first and second day after the surgical procedure, and during the first follow-up with the oncological surgeon.

Additionally, the investigators collected samples of cancerous colon mucosa from 10 participants for the attempt to isolate F. nucleatum and P. gingivalis using the quantitative culture method.

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer, scheduled for surgical treatment
* consent to participate

Additional inclusion Criteria fot the control group:

* fiilled questionnaire
* Recorded CRP results at the first examination, after surgery, and at the first follow-up examination.

Exclusion Criteria:

* under 18 years old
* periodontal treatment in the past 12 months
* antibiotic therapy in the last 3 months
* edentulism
* advanced stage cancer, scheduled for palliative care
* chemotherapy or radiotherapy prior to surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
CRP levels | From the enrollment to the date of first documented progression at 16 weeks
  Measurement of CRP levels in the blood of patients with colorectal cancer at the first examination by the oncological surgeon, on the first and second day after colon resection, and at the first follow-up examination by the oncological surgeon.
The proportion of Fusobacterium nucleatum and Porphyromonas gingivalis | From the first dental exam to the resective colon surgery at 2 weeks
  Using quantitative culture for detection of periodontal bacteria Fusobacterium nucleatum and Porphyromonas gingivalis in the cancer altered intestinal musoca and comparing it with the status in the periodontal pocket

CONTACTS AND LOCATIONS:
Overall Officials: Rok Schara, associate professor, doctor of dental medicine, Study Director — University Medical Cneter Ljubljana, Division of Stomatology, Center of oral disease and periodontology,
Locations (1):
- University Medical Center Ljubljana, Division of stomatology, Center for oral disease and periodontology, Ljubljana, Slovenija, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
sex, age, clinical diagnosis and location of colorectal cancer, histological diagnosis of the cancer, stage of cancer, BMI, Smoker or not, possible concomitant systemic diseases
Supporting Information: Study Protocol, SAP, CSR